CLINICAL TRIAL: NCT00878397
Title: Evaluating the Impact of Delivering Long Lasting Insecticide Nets Through Schools on Household Access and the Health of School Children in North Eastern Kenya
Brief Title: Impact of School-based Delivery of Long Lasting Insecticide Nets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Principal Investigator, Simon Brooker, Professor of Epidemiology, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5482
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Malaria
Keywords: malaria; long lasting insecticide nets; anaemia; schools
MeSH Terms: conditions — Malaria; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Free distribution of long lasting insecticide nets to school children and their younger siblings
  Interventions: Device: School-based delivery of long lasting insecticide nets
- 2 (Experimental): No school-based delivery of long lasting insecticide nets in the first year, followed by free delivery in the second year
  Interventions: Device: School-based delivery of long lasting insecticide nets

INTERVENTIONS:
Device: School-based delivery of long lasting insecticide nets — Free distribution of long lasting insecticide nets to school children and their younger siblings

SUMMARY:
Insecticide-treated nets (ITNs), and more recently long lasting insecticide nets (LLINs), have been shown to effectively protect those groups most biologically vulnerable to the burden of malaria across Africa. However, achieving universal coverage, especially in poor and remote areas, has proved a particular challenge and there remains a need to explore alternative delivery mechanisms. The recent introduction of universal primary education in Kenya has meant that even the poorest households are sending at least one child to school, providing a complementary, potentially equitable, mechanism through which to distribute LLINs. The delivery of LLINs through schools will be piloted by Population Services International in schools situated along the Tana River in North Eastern Kenya. This proposal seeks to evaluate the impact of this programme on both household use of school donated, free LLINs and the health of schoolchildren. The study hypothesis is that the free delivery of long lasting insecticide nets (LLINs) through schools will increase household LLIN coverage among younger siblings not enrolled in school and will reduce rates of malaria infection and anaemia among school children. The study will be an impact evaluation of a programme delivering LLINs through schools, which is to be implemented by Population Services International (PSI)-Kenya. The programme will be implemented in 50 schools and due to PSI-Kenya's roll out, the programme will be phased in over two years. will be phased in over two years. The 50 schools will be randomly divided into two groups, the first 25 schools will receive LLINs in 2009 and the second group will receive them in 2010. In each school, five households will be randomly selected and household surveys will be conducted to collect information on household net use and household demographic and socio-economic status. School health surveys will be completed at the end of the programme to assess programme impact on malaria infection and anaemia.

ELIGIBILITY:
Inclusion Criteria:

* Pupil enrolled at participating schools in standards 1-7;
* Provision of informed consent from parent or guardian; AND
* Provision of assent by student.

Exclusion Criteria:

* Non-provision of informed consent; OR
* Pupils unwilling to participate in the study.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5113 (Actual)
Dates: Start 2009-05; Primary Completion 2010-07 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Anaemia | 2 years

SECONDARY OUTCOMES:
Household coverage and use of long lasting insecticide nets | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Simon Brooker, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine / KEMRI-Wellcome Trust Programme
Locations (1):
- KEMRI-Wellcome Trust Programme, Nairobi, Kenya